CLINICAL TRIAL: NCT03535077
Title: Assessing Tissue Remodeling in the Skin Using Skin Fluorescence Imaging (SFI)
Brief Title: Assessing Tissue Remodeling in the Skin Using SFI (Skin Fluorescence Imaging)
Status: Completed | Type: Observational
Sponsor: Orlucent, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SFI 001
Record Dates: First submitted 2018-02-14; First posted 2018-05-24 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Skin Lesion; Melanoma (Skin); Mole
Keywords: Melanoma; Nevus; Mole; Atypical Nevi
MeSH Terms: conditions — Melanoma; Nevus; Dysplastic Nevus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicious Nevi undergoing biopsy: Subject with suspicious Nevi undergoing biopsy per SOC
  Interventions: Other: Diagnostic Test

INTERVENTIONS:
Other: Diagnostic Test — Imaging of the suspicious lesion after application of ORL-1 dye prior to biopsy
  Other Names: SFI 001 Imaging

SUMMARY:
The goal of the SFI is to provide non-invasive information about tissue remodeling occurring during melanocytic transition and atypia development in the skin

DETAILED DESCRIPTION:
The goal of the SFI is to provide non-invasive information about tissue remodeling occurring during melanocytic transition and atypia development in the skin. SFI analyzes the topical staining of the skin surface using the ORL-1 dye to reveal the presence of remodeling in the skin, together with the visible feature characteristics. The system provides a biometric score corresponding to the dye staining, a structural score, and a composite SFI score to quantify the presence of tissue remodeling and the process of melanocytic transition in the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a pigmented skin lesion recommended for a skin biopsy.
2. A lesion that is accessible to the imaging device, with at least 1 cm of skin around the lesion that is accessible to the MDS.
3. At least 21 years old.
4. Written, signed, and dated informed consent
5. Scheduled for a primary excision/biopsy as part of the clinics SOC.

Exclusion Criteria:

1. Lesion is less than 1 centimeter from the eyes.
2. Lesion is on the palms of the hands or soles of the feet.
3. Mucosal lesion.
4. Ulcerated lesion.
5. Subject is pregnant or planning to become pregnant during the study period.
6. Patients who are mentally or physically unable to comply with all aspects of the study.
7. Any subject undergoing chemotherapy.
8. Any lesion that has been treated with local anesthesia such as lidocaine prior to enrollment that would confound study results.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll subjects being evaluated for suspicious moles/nevi and who will be scheduled to undergo a biopsy of the mole/nevus as part of the physicians standard plan of care.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation | 1 day
  To identify histological features that correlate with the imaging features captured using SFI

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Shachaf, PhD, Study Director — President
Locations (6):
- United States (6):
  - Center for Dermatology Clinical Research, Inc, Fremont, California
  - UCI Center for Clinical Research, Irvine, California
  - Divya Railan, Md, Faad, Menlo Park, California
  - Quest Dermatology Research, Northridge, California
  - Solano Dermatology Associates, Vallejo, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Undecided